CLINICAL TRIAL: NCT06509633
Title: Effects of Pain Neuroscience Education and Standard Rehabilitation Regime in Patients of Carpal Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/01113
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Wrist Injuries; Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; Compression; Pain neuroscience education; Median nerve
MeSH Terms: conditions — Wrist Injuries; Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience education and Standard Rehabilitation regime (Experimental): Patients will get standard treatment of CTS, which is nerve gliding, stretchings of forearm and wrist muscles and wrist mobilization along with pain neuroscience education.
  Interventions: Other: Pain Neuroscience education and standard rehabilitation regime
- standard Rehabilitation regime (Active Comparator): Patient will get only nerve gliding and wrist forearm muscle stretching exercises.
  Interventions: Other: standard Rehabilitation regime

INTERVENTIONS:
Other: Pain Neuroscience education and standard rehabilitation regime — Median nerve gliding exercises, wrist and forearm muscle stretches, wrist mobilizations and finger joint mobilizations
  Other Names: Standard Rehabilitation regime
  Arms: Pain Neuroscience education and Standard Rehabilitation regime
Other: standard Rehabilitation regime — standard Rehabilitation regime
  Arms: standard Rehabilitation regime

SUMMARY:
The aim of this study is to check the effects of Pain Neuroscience education and standard rehabilitation regime in patients of carpal tunnel syndrome.

DETAILED DESCRIPTION:
In 2017 a stud assessed effectiveness of standard conservative protocol of CTS and nerve mobilization along with and without PNE and documented that standard conservative care seems to be the most appropriate option for pain relief, although neuroscience education might be a complementary option to accelerate recovery of function. More high-quality research is still necessary to determine its effectiveness and the subgroups of patients who may respond better to this treatment.

In 2019 a study was done to assess the effect of PNE and standard rehabilitation exercises on the 41 patients of CTS. The experimenting group was given one session of PNE plus exercises and the control group was given exercise therapy only. Patients were randomly allocated and double blinded. The analysis of study showed better results with experimental group rather than control group.

Many studies have found the effects of standard rehabilitation of Carpal Tunnel syndrome and their results in controlling pain and dysfunction. However as per researchers' knowledge little literature is available on effects of pain neuroscience education and standard rehabilitation regime in carpal tunnel syndrome. Therefore, this study6 is going to determine the effects of effectiveness of Pain Neuroscience education and standard rehabilitation regime in patients of carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age between 20_40 years old.
* Medical diagnosis of moderate to severe CTS.
* Symptoms of CTS since 1month
* Unilateral or bilateral symptoms
* Availability and access to the hospital.

Exclusion Criteria:

* Inability to understand instructions, neurological conditions of the central nervous system (e.g. stroke, spinal cord injury)
* Patients on treatment with alternative therapies
* Previous participation in a research program
* Previous surgery on the affected upper limb

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Carpal Tunnel syndrome is prevalent in female housewives and computer users.
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rate scale (NPRS) | 4th week
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS) | 4th week
  The Pain Catastrophizing Scale (PCS) was used to measure catastrophic thinking in response to pain through 13 statements with four possible options, from 1 "not at all" to 4 "all the time".

OTHER OUTCOMES:
Boston Carpal Tunnel Questionnaire (BCTQ) | 4th week
  BCTQmeasures self reported functional status and severity of symptom. The BCTQ-SSS consists of 11 questions, each question provides 5 response choices, from 1 (no symptoms) to 5 (most severe/often).
Goniometer | 4th week
  The range of motions like flexion extension radial deviation and ulnar deviation of wrist will be measured by Goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Saba khan, Principal Investigator — Riphah International University
Locations (1):
- Absaar medical center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Werner RA, Andary M. Electrodiagnostic evaluation of carpal tunnel syndrome. Muscle Nerve. 2011 Oct;44(4):597-607. doi: 10.1002/mus.22208. PMID 21922474
- [Background] Genova A, Dix O, Saefan A, Thakur M, Hassan A. Carpal Tunnel Syndrome: A Review of Literature. Cureus. 2020 Mar 19;12(3):e7333. doi: 10.7759/cureus.7333. PMID 32313774
- [Background] Nunez-Cortes R, Espinoza-Ordonez C, Pommer PP, Horment-Lara G, Perez-Alenda S, Cruz-Montecinos C. A single preoperative pain neuroscience education: Is it an effective strategy for patients with carpal tunnel syndrome? Med Hypotheses. 2019 May;126:46-50. doi: 10.1016/j.mehy.2019.03.013. Epub 2019 Mar 22. PMID 31010499
- [Background] Nunez-Cortes R, Cruz-Montecinos C, Torreblanca-Vargas S, Tapia C, Gutierrez-Jimenez M, Torres-Gangas P, Calatayud J, Perez-Alenda S. Effectiveness of adding pain neuroscience education to telerehabilitation in patients with carpal tunnel syndrome: A randomized controlled trial. Musculoskelet Sci Pract. 2023 Oct;67:102835. doi: 10.1016/j.msksp.2023.102835. Epub 2023 Jul 28. PMID 37572618
- [Background] Ballestero-Perez R, Plaza-Manzano G, Urraca-Gesto A, Romo-Romo F, Atin-Arratibel MLA, Pecos-Martin D, Gallego-Izquierdo T, Romero-Franco N. Effectiveness of Nerve Gliding Exercises on Carpal Tunnel Syndrome: A Systematic Review. J Manipulative Physiol Ther. 2017 Jan;40(1):50-59. doi: 10.1016/j.jmpt.2016.10.004. Epub 2016 Nov 11. PMID 27842937
- [Background] Bulow K, Lindberg K, Vaegter HB, Juhl CB. Effectiveness of Pain Neurophysiology Education on Musculoskeletal Pain: A Systematic Review and Meta-Analysis. Pain Med. 2021 Apr 20;22(4):891-904. doi: 10.1093/pm/pnaa484. PMID 33764394
- [Background] Louw A, Puentedura EJ, Zimney K, Schmidt S. Know Pain, Know Gain? A Perspective on Pain Neuroscience Education in Physical Therapy. J Orthop Sports Phys Ther. 2016 Mar;46(3):131-4. doi: 10.2519/jospt.2016.0602. PMID 26928735
- [Background] Ziegler AM, Minkalis AL, Langdon ER, Vining R. Learning the neurobiology of pain: A scoping review of pain education from an instructional design perspective. Patient Educ Couns. 2022 Jun;105(6):1379-1401. doi: 10.1016/j.pec.2021.09.021. Epub 2021 Sep 14. PMID 34579995
- [Background] Lopez-de-Uralde-Villanueva I, Fernandez-de-Las-Penas C, Cleland JA, Cook C, de-la-Llave-Rincon AI, Valera-Calero JA, Plaza-Manzano G. Minimal Clinically Important Differences in Hand Pain Intensity (Numerical Pain Rate Scale) and Related-Function (Boston Carpal Tunnel Questionnaire) in Women With Carpal Tunnel Syndrome. Arch Phys Med Rehabil. 2024 Jan;105(1):67-74. doi: 10.1016/j.apmr.2023.07.018. Epub 2023 Aug 13. PMID 37582474
- [Background] Sullivan MJ, Bishop SR, Pivik J. The pain catastrophizing scale: development and validation. Psychological assessment. 1995;7(4):524.
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050